CLINICAL TRIAL: NCT04644679
Title: 48-hour Versus 7-day Monitoring for the Detection of Atrial Fibrillation in Patients with Cryptogenic Stroke
Brief Title: Monitoring Strategies for the Detection of Atrial Fibrillation in Patients with Cryptogenic Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment rate
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, EMILIANO ROSSI, MD, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5767
Record Dates: First submitted 2020-09-30; First posted 2020-11-25 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2020-11

CONDITIONS: Stroke; Atrial Fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 48-hr (Active Comparator): 48-hr electrocardiographic monitoring
  Interventions: Diagnostic Test: 48-hr electrocardiographic monitoring
- 7-day (Experimental): 7-day electrocardiographic monitoring
  Interventions: Diagnostic Test: 7-day electrocardiographic monitoring

INTERVENTIONS:
Diagnostic Test: 7-day electrocardiographic monitoring — 7-day external electrocardiographic monitoring
  Arms: 7-day
Diagnostic Test: 48-hr electrocardiographic monitoring — 48-hr external electrocardiographic monitoring
  Arms: 48-hr

SUMMARY:
Randomized clinical trial comparing two monitoring strategies, the use of a 48-hour Holter (routine care branch) and an event recorder for 7 days (intervention branch).

Patients admitted for cryptogenic stroke will be included. Enrollment and randomization of patients will be carried out during the index case hospitalization, while follow-up will be done on an outpatient basis until day 7.

DETAILED DESCRIPTION:
Once the diagnose of cryptogenic stroke have been carried out, informed consent will be taken and participants will be randomized to 48-hour monitoring arm or 7-day monitoring arm, followed by discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have studies that classify stroke or TIA as cryptogenic and who can carry out monitoring for 48 hours or 7 days will be included.
* Age ≥ 18 years

Exclusion criteria

* History of atrial fibrillation (or atrial flutter) documented.
* Patients who already have an event recorder in place, permanent pacemaker, or implantable cardioverter-defibrillator
* Evidence of lacunar infarction.
* Hemorrhagic stroke
* Patient for palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation | 7 days
  Detection of one episode of atrial fibrillation or atrial flutter >30 seconds up to 7 days

SECONDARY OUTCOMES:
Supraventricular arrhythmia | 7 days
  Count of beats per day of non-sustained irregular atrial tachyarrhythmia or supraventricular extrasystoles up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Maid, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, C.a.b.a, Argentina

IPD SHARING:
Plan to Share IPD: No